CLINICAL TRIAL: NCT06976593
Title: Analysis of Muscle Oxygen Saturation and Functional Variables During Physical Performance Tests in Breast Cancer Survivors
Brief Title: Muscle Oxygen Saturation and Functional Capacity in Breast Cancer Survivors
Status: Not yet recruiting | Type: Observational
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Investigator, University of Extremadura
Other Study IDs: 050525
Record Dates: First submitted 2025-05-05; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Survivorship; Muscle Oxygenation; Near-infrared Spectroscopy; Exercise; Quality of Life; Functional Capacity; Hormonal Therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hormonal Therapy Only: Participants who received only hormonal therapy following breast cancer treatment.
  Interventions: Diagnostic Test: Functional Exercise Testing and Muscle Oxygen Saturation Measurement
- Hormonal Therapy + Chemotherapy: Participants who received both hormonal therapy and chemotherapy.
  Interventions: Diagnostic Test: Functional Exercise Testing and Muscle Oxygen Saturation Measurement

INTERVENTIONS:
Diagnostic Test: Functional Exercise Testing and Muscle Oxygen Saturation Measurement — Participants will complete three physical performance tests: (1) the 6-Minute Walk Test (6MWT), (2) the 30-Second Sit-to-Stand Test, and (3) a submaximal treadmill test. Muscle oxygen saturation (SmO2) will be continuously monitored during the tests using near-infrared spectroscopy (NIRS) devices placed on the intercostal, quadriceps, and triceps surae muscles. Additional variables such as heart rate, perceived exertion, respiratory pressures, pulmonary function, and fatigue will be assessed during or after the tests.

SUMMARY:
This cross-sectional observational study aims to assess muscle oxygen saturation (SmO2) in the intercostal, quadriceps, and triceps surae muscles using near-infrared spectroscopy (NIRS) during functional exercise tests in breast cancer survivors. Participants will be grouped based on their previous cancer treatment: hormonal therapy only or hormonal therapy combined with chemotherapy. Functional performance will be evaluated through the 6-Minute Walk Test, 30-Second Sit-to-Stand Test, and a submaximal treadmill test. The study will analyze differences in muscle oxygenation and performance between groups and explore associations with other functional and clinical parameters.

DETAILED DESCRIPTION:
This study focuses on evaluating muscle oxygen saturation and physical performance in women who have survived breast cancer. Cancer treatments such as chemotherapy and hormonal therapy can lead to systemic effects, including muscular deconditioning, fatigue, and reduced cardiorespiratory capacity. Near-infrared spectroscopy (NIRS) offers a non-invasive means of assessing SmO2 in real-time, providing insight into oxygen delivery and utilization during exercise.

Participants will undergo three functional tests: the 6-Minute Walk Test, the 30-Second Sit-to-Stand Test, and a submaximal treadmill test. Muscle oxygenation will be measured in three key muscle groups before, during, and after each task. Additional outcomes include functional test performance, respiratory strength, pulmonary function, fatigue perception, and quality of life questionnaires. This study will explore whether prior cancer treatment protocols affect muscle oxygenation and physical function differently, and may inform future rehabilitation strategies tailored to breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 to 70 years
* Clinical history of breast cancer treatment (at least 6 months prior)
* Completed primary cancer treatment
* Ability to perform physical tests
* Signed informed consent

Exclusion Criteria:

* Recurrence or metastasis
* Severe cardiopulmonary or musculoskeletal disease
* Neurological or cognitive limitations
* Ongoing oncological treatment

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of women aged 30 to 70 years who have completed treatment for breast cancer. Participants are recruited from outpatient oncology clinics and cancer survivor support groups in the region of Extremadura, Spain. All participants are categorized into two groups based on their treatment history: those who received hormonal therapy only and those who received both hormonal therapy and chemotherapy. All subjects must be able to perform physical tests and attend a single evaluation session.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Muscle oxygen saturation (%) | Within a single assessment session (~1 hour)
  Measured via NIRS in intercostal, quadriceps, and triceps surae muscles during three functional tests (6MWT, 30CST, treadmill)

SECONDARY OUTCOMES:
Distance covered in the 6-Minute Walk Test (meters) | During and immediately after functional assessment session
Number of repetitions in the 30-Second Sit-to-Stand Test | During and immediately after functional assessment session
Maximal heart rate and recovery rate during treadmill test | During and immediately after functional assessment session
Lower limb fatigue and perceived exertion (Borg scale) | During and immediately after functional assessment session
  0-10 points. 0: no perceived effort 10: maximum perceived effort
Maximal inspiratory pressures (Pimax) | During and immediately after functional assessment session
Pulmonary function (FEV1/FEV6 ratio using Vitalograph® COPD-6) | During and immediately after functional assessment session
Quality of life (EORTC QLQ-C30) European Organisation for Research and Treatment of Cancer | During and immediately after functional assessment session
Maximal expiratory pressures (Pemax) | During and immediately after functional assessment session
Quality of life (BR23) | During and immediately after functional assessment session

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Mecina y Ciencias de la Salud, Badajoz, Spain